CLINICAL TRIAL: NCT02949310
Title: Effectiveness of Nefopam in Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Clinical professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Nefo-TM & MRM
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Breast Neoplasm Malignant Primary
MeSH Terms: interventions — Nefopam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Control (Placebo Comparator): Placebo use instead of nefopam
  Interventions: Drug: Normal Saline
- Nefopam (Experimental): Intraoperative use of nefopam 40 mg
  Interventions: Drug: Nefopam

INTERVENTIONS:
Drug: Nefopam
  Arms: Nefopam
Drug: Normal Saline
  Arms: Control

SUMMARY:
Breast cancer surgery is known to cause severe acute postoperative pain, which can persist for a long time. The investigators administered nefopam preventively to patients undergoing total mastectomy or modified radical mastectomy with axillary lymph node dissection or sentinel lymph node biopsy, and evaluated its efficacy on acute and chronic postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Total mastectomy
* Modified radical mastectomy
* Nipple-sparing mastectomy
* American Society of Anesthesiologists physical status I or II
* Postoperative use of intravenous patient-controlled analgesia

Exclusion Criteria:

* Chronic analgesia medication
* Pregnancy
* Lactating women
* Previous operation history due to breast cancer
* Cooperation with other surgery
* Contraindication of nefopam

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change of cumulative analgesia volume infused via intravenous patient-controlled analgesia device | At postoperative 4 hour, 24 hour, 48 hour, 72 hour, 10 day, and 3 month

SECONDARY OUTCOMES:
Change of numerical rating scale for postoperative pain | At postoperative 4 hour, 24 hour, 48 hour, 72 hour, 10 day, and 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea